CLINICAL TRIAL: NCT04309552
Title: A Phase-I Trial for Simultaneous Imaging of Tumor Hypoxia and Proliferation in Patients With Treatment- Naïve High-Grade Glioma
Brief Title: Tumor Hypoxia and Proliferation in Patients With High-Grade Glioma
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The study team would like to implement an amendment to the protocol with the corresponding IRB before continuing with recruitment.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: William Rhodes Center for Glioblastoma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-02021553
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — fluoromisonidazole

STUDY DESIGN:
Intervention Model Description: Single center, prospective, non-randomized trial of 30 newly diagnosed patients with suspected HGG undergoing surgical planning will be enrolled to undergo combined FMISO/FLT PET at baseline. Blood samples will be drawn during PET acquisition. Preoperatively FMISO/FLT PET data will be used for intraoperative neuro-navigation and targeted sampling of PET avid tumor subregions prior to tumor excision. Paraffin blocks will be analyzed with immuno-histochemistry and in situ hybridization. Longitudinal clinical data will be collected from the medical record for standard of care visits to the oncology and surgical clinics. Imaging data from research scans will be correlated with time to progression, progression-free survival at 9 months, and overall survival (OS) at 1 year post baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- High Grade Glioma (HGG) (Experimental): Thirty newly diagnosed treatment-naïve subjects with suspected HGG based on clinical presentation and MRI findings and undergoing surgical planning will be accrued in this study.
  Interventions: Drug: 18F-FMISO PET; Drug: 18F-FLT PET

INTERVENTIONS:
Drug: 18F-FMISO PET — Suspected HGG subjects will undergo combined FMISO/FLT dyn-PET at baseline as part of surgical planning. Dyn-PET images will be acquired with staggered FMISO/FLT injections using a lag time of 50 minutes. Preoperatively FMISO/FLT dyn-PET data will be used for intraoperative neuro-navigation and targeted sampling of PET avid tumor subregions prior to tumor excision. Paraffin blocks will be analyzed with immuno-histochemistry and in situ hybridization for HIF-1α, Ki-67, VEGF, EGFR, IDH, and pimonidazole, as well as TERT. FMISO-PET uptake rate, k3, (surrogate for hypoxia) and FLT-PET influx rate, Ki (surrogate for proliferation) will be correlated with time to progression, progression-free survival at 9 months, and overall survival (OS) at 1 year.
  Other Names: 18F-Fluoromisonidazole
Drug: 18F-FLT PET — Suspected HGG subjects will undergo combined FMISO/FLT dyn-PET at baseline as part of surgical planning. Dyn-PET images will be acquired with staggered FMISO/FLT injections using a lag time of 50 minutes. Preoperatively FMISO/FLT dyn-PET data will be used for intraoperative neuro-navigation and targeted sampling of PET avid tumor subregions prior to tumor excision. Paraffin blocks will be analyzed with immuno-histochemistry and in situ hybridization for HIF-1α, Ki-67, VEGF, EGFR, IDH, and pimonidazole, as well as TERT. FMISO-PET uptake rate, k3, (surrogate for hypoxia) and FLT-PET influx rate, Ki (surrogate for proliferation) will be correlated with time to progression, progression-free survival at 9 months, and overall survival (OS) at 1 year.
  Other Names: 3'-deoxy- 3'[(18)F]-fluorothymidine

SUMMARY:
This is a pilot study to assess a new methodology developed for High Grade Glioma (HGG). FMISO PET (Fluoromisonidazole-PET) allows researchers to study whether tumor cells lack oxygen (hypoxia). FLT PET (Fluorodeoxythymidine-PET) allows researchers to study the increase in the number of cells as a result of cell growth and cell division (proliferation). Tumors that have low oxygen levels and/or are dividing fast shall resist to standard cancer treatment. The study will compare FMISO PET and FLT PET imaging techniques with molecular biomarkers of hypoxia, angiogenesis, and cellular proliferation in tissue. proliferation).This information could help researchers develop new treatment techniques to better treat cancer.

DETAILED DESCRIPTION:
This is a pilot study to assess a novel methodology recently developed to simultaneously image tumor hypoxia and proliferation by means of simultaneous FMISO and FLT PET acquisition. FMISO (18F-Fluoromisonidazole) PET is a non-invasive method for detecting tumor hypoxia in solid tumors. FLT (3'-deoxy-3'[(18)F]-fluorothymidine) PET is a non-invasive method to image Cell proliferation rate. Imaging of tumor hypoxia and proliferation with FMISO and FLT PET respectively are two very well established techniques in in high-grade glioma. The long-term goal of this proposal is to establish clinically robust methodology to simultaneously image multiple tumor hallmarks. The central hypothesis is that combined information from multiple tumor hallmarks will offer complementary information about the underlying physiological processes, and will yield synergistic prognostic and predictive values. The rationale is that these findings will enhance the understanding of the underlying biology and pathophysiology, and will open new therapeutic strategies to target radioresistant and highly aggressive regions within the tumor, as well as aiding in the development of imaging theragnostics. The method used in this proposal is based on our previous work on simultaneous imaging of FMISO/FLT PET, and is facilitated by prior knowledge of the tissue pharmacokinetics, and an ability to distinguish the two radiotracers fractions in blood by thin-layer chromatography (TLC). The study will compare FMISO and FLT imaging findings with those from molecular biomarkers of hypoxia, angiogenesis, and cellular proliferation in tissue.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Documentation of a suspected HGG diagnosis based on clinical and MRI findings

Exclusion Criteria:

* Pregnant or breastfeeding
* Contraindications to receiving Positron Emission Tomography (PET) imaging (e.g. claustrophobia)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Quantitation of tumor hypoxia (FMISO) by measuring Dyn PET | 1 year
  Simultaneous quantitation of tumor hypoxia (FMISO): Dyn-PET data will be acquired with staggered FMISO/FLT injections and then the two radiotracer signals will be deconvolved using our novel pharmacokinetics modeling approach (Sections D2, D3, and D4 of Preliminary Data)
Quantitation of proliferation (FLT) by measuring Dyn PET | 1 year
  Simultaneous quantitation of proliferation (FLT): Dyn-PET data will be acquired with staggered FMISO/FLT injections and then the two radiotracer signals will be deconvolved using our novel pharmacokinetics modeling approach (Sections D2, D3, and D4 of Preliminary Data)

SECONDARY OUTCOMES:
FMISO/FLT PET Metrics and Molecular Biomarkers of Tissue Hypoxia, Tissue Angiogenesis, and Tissue Proliferation | 1 year
  FMISO/FLT images will be used for intraoperative neuro-navigation and targeted sampling of FMISO and FLT avid tumor subregions prior to tumor excision. PET metrics will be correlated with immuno-histochemistry (IHC) analyses for HIF-1α, Ki-67, VEGF, EGFR, IDH1, and pimonidazole, as well as molecular analyses of TERT promoter mutation status. Results will be based on a composite score from all measurements. These markers contribute to disease progression in HGG.

CONTACTS AND LOCATIONS:
Overall Officials: Sadek Nehmeh, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No